CLINICAL TRIAL: NCT03346954
Title: Impact of [11C]-Methionine PET/MRI in the Detection of Pituitary Adenomas Secreting ACTH and Causing Cushing's Disease
Acronym: IMPEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0167; 2017-002721-38 (EudraCT Number)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2020-11

CONDITIONS: Cushing's Disease
Keywords: : Cushing's disease, [11C]-Methionine PET/MRI, Sensitivity
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Cushing's disease (Experimental): Implementation of [11C]-Methionine PET/MRI
  Interventions: Other: [11C]-Methionine PET/MRI

INTERVENTIONS:
Other: [11C]-Methionine PET/MRI — Implementation [11C]-Methionine PET/MRI performed for each patient in one place (department of nuclear medicine of the Hospices Civils de Lyon). The [11C]-Methionine PET/MRI will be performed after a pituitary MRI and before a transsphenoidal surgery.

SUMMARY:
Cushing's disease is characterized by the existence of a benign pituitary tumor developed from corticotropic cells responsible for excessive ACTH secretion. This results in hypercorticism causing high morbidity and mortality and severely impairing quality of life. The etiological diagnosis is based on Magnetic Resonance Imaging (MRI). However, pituitary MRI revealed a pituitary tumor in only 60% of patients. The diagnostic procedure is complicated by the existence of extra pituitary tumors responsible for ACTH ectopic secretion. This rare etiology imposes, in the absence of typical pituitary image, the realization of catheterization of the lower petrosal sinuses. Treatment of Cushing's disease is based on transsphenoidal surgical management, even in the absence of a formal MRI image, if pituitary origin is confirmed by the catheterization. Although pituitary surgery without identified target is part of French recommendations, this surgery is associated with a high risk of failure and morbidity. Optimization of the management of patients' with Cushing's disease thus requires the improvement of the diagnostic methods.

Hypothesis of our study is that [11C] MET MRI-PET may be performed as a first-line MRI for suspected Cushing's disease and may limit indications for catheterization of lower petrosal sinuses. Its localizing value should also make it possible to improve the surgical results with a better identification of the adenoma

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or over
* Patient with a diagnosed Cushing's disease according to the French "protocole national de diagnostic et de soins (PNDS)"
* Patient who underwent a MRI pituitary for diagnostic purposes
* Patient who have undergone catheterization of the lower petrosal sinuses (if MRI does not detect pituitary adenoma) and have a result in favor of a central secretion of ACTH
* Patient having an indication of surgical excision of the adenoma
* Patient with a micro-adenoma (less than 1 cm in diameter) if the tumor is visualized on MRI
* Patient for which informed and written consent to participate has been obtained.

Exclusion Criteria:

* - Patient participating in another study
* Patient with a pituitary macro-adenoma with visual impairment
* Patient with ACTH-dependent Cushing's syndrome secondary to ectopic ACTH secretion
* Patient with recurrence and / or history of pituitary adenoma excision
* Patient with a contraindication to pituitary surgery or general anesthesia
* Pregnant woman, breastfeeding or old enough to have children but without effective recognized contraception
* Contra-indication to the realization of an MRI: permanently fixed metal parts (pacemaker, cerebral clip, cephalic end piercing, cochlear implant, pin or screw for recent bone fracture, dental equipment, metal splinters), claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of [11C]-Methionine PET/MRI | Within 3 months and 3 weeks after inclusion
  Sensitivity of [11C]-Methionine PET/MRI to correctly localizes the pituitary corticotropic adenoma in comparison with the sensitivity of the pituitary MRI. The gold standard being the localization defined by anatomopathological analysis on operative resection.

SECONDARY OUTCOMES:
False negatives and false positives description | Within 3 months and 3 weeks after inclusion
  Description of false negatives and false positives [11C]-Methionine PET/MRI to identify and localize the microadenoma. Characteristics of unidentified adenomas will be described using: volume, localization, type of fixation
Description of identified microadenomas | Within 3 months and 3 weeks months after inclusion
  Proportion of microadenomas identified by the [11C]-Methionine PET/MRI as a function of the degree of aggressiveness of the adenoma, evaluated by the number of mitoses, the level of expression of Ki67 and p53.
Comparison of [11C]-Methionine PET/MRI and pituitary MRI | Within 3 months and 3 weeks months after inclusion
  Study of the concordance between the results of [11C]-Methionine PET/MRI and pituitary MRI

CONTACTS AND LOCATIONS:
Overall Officials: BOURNAUD Claire, MD, Study Director — Hospices Civils de Lyon
Locations (1):
- Service de Médecine Nucléaire - Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flaus A, Levigoureux E, Haesebaert J, Briet C, Castinetti F, Cristante J, Drui D, Germain N, Maione L, Illouz F, Sonnet E, Tauveron I, Merida I, Lancelot S, Costes N, Vasiljevic A, Marchand L, Rode S, Bertholon-Gregoire M, Criton G, Lapras V, Cotton F, Jouanneau E, Bournaud C, Raverot G. Prospective Multicenter Evaluation of [11C]Methionine PET/MRI Sensitivity Compared with MRI for Localizing Small Pituitary Neuroendocrine Tumor or Pituitary Adenoma in Cushing Disease. J Nucl Med. 2025 Oct 1;66(10):1575-1580. doi: 10.2967/jnumed.124.269392. PMID 40841148